CLINICAL TRIAL: NCT06995742
Title: Effect of ANNE One-Wellue Device Array Use on Staff Bedside Vital Sign Measurement Activity: A Randomized Controlled Trial
Brief Title: Effect of ANNE One-Wellue Device Array Use on Staff Bedside Vital Sign Measurement Activity
Acronym: ANNE One TMRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Minnesota Medical School/University of Minnesota Foundation (Unknown); Sibel Health Inc. (Industry)
Responsible Party: Principal Investigator, Gregory Randall Smith Jr, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00219340; 2023 Dixon Translational Grant (Other Grant/Funding Number: Northwestern University Clinical and Translational Sciences Institute)
Record Dates: First submitted 2025-04-29; First posted 2025-05-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Vital Sign Evaluation; Vital Sign Monitoring; Sleep Quality; Provider Behavior; Patient Satisfaction
Keywords: time motion study; vital signs; sleep quality; inpatient sleep; wireless device; patient satisfaction
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention--Device Array Use (Experimental): Inpatients will wear the ANNE One device array for obtainment of vital sign assessments.
  Interventions: Device: Device Array Use
- Control--Routine Vital Sign Obtainment (Active Comparator): Inpatients will have vital signs determined by routine practice, using any other standard of care-accepted method or device.
  Interventions: Device: Routine Vital Sign Measurement

INTERVENTIONS:
Device: Device Array Use — Study participants assigned to the intervention study arm will wear a wireless Bluetooth capable vital sign detection array, with one device externally worn on each of their chest, one finger, and one arm, with healthcare providers using an additional oral temperature probe.
  Arms: Intervention--Device Array Use
Device: Routine Vital Sign Measurement — Study participants randomized to the control arm will have their vital signs obtained by routine means, without use of the wireless vital sign device array.
  Arms: Control--Routine Vital Sign Obtainment

SUMMARY:
Randomized controlled trial of a time motion study of time spent obtaining and charting vital signs for inpatients, comparing use of a wireless Bluetooth vital sign array as intervention versus routine vital sign obtainment activity on a general medical floor.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients admitted to Northwestern Memorial Hospital, Feinberg Unit 16 West.

Exclusion Criteria:

* Primary language other than English, under isolation status, pregnant patients, prisoners, employees or students of the hospital or Northwestern University.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time Motion Assessment of Time Spent Obtaining and Recording Vital Signs | Number of seconds spent obtaining and charting vital signs is obtained at 8a daily, for maximum of three days for each study participant, and are added together to equal the total time spent on vital sign assessment.
  The number of seconds spent by a healthcare provider obtaining and charting vital signs will be witnessed and recorded by a research staff member.

SECONDARY OUTCOMES:
Sleep Quality of Inpatient Study Participants | Survey conducted 24-72 hours after enrolment.
  Sleep quality will be determined by use of the Potential Hospital Sleep Disruptions and Noises Questionnaire survey, administered to study participants after a night of study enrolment. The survey scores sleep quality from 1 to 5 with 1 signifying no disruption and 5 signifying extreme disruption.
Patient Satisfaction with Inpatient Sleep Quality | Survey sent within a week of hospital discharge and collected within the subsequent thirty days.
  Question 8, "During this hospital stay, how often were you able to get the rest you needed?" of the Hospital Consumer Assessment of Healthcare Providers and Systems post-discharge questionnaire will be collected for study participants. Survey responses include: never, sometimes, usually, always.
Healthcare Provider Experience with the Vital Sign Device Array | The electronic survey will be administered twice during the study. Each survey will take approximately ten minutes to complete.
  Healthcare providers who use the device array will be surveyed with a Technology Acceptance Method survey to assess usability of the device array.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory (Randy) R Smith Jr, MD MS, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (2):
- United States (2):
  - Feinberg 16 West, Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No